CLINICAL TRIAL: NCT02496351
Title: Transcutaneous Electrical Nerve Stimulation (TENS) for Phantom Limb Pain Prevention Following Arteriopathic Major Amputation: Clinical Trial
Brief Title: TENS for Phantom Limb Pain Prevention Following Major Amputation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Barbara Bodega, MD, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 161976BBM
Record Dates: First submitted 2015-07-09; First posted 2015-07-14 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-06

CONDITIONS: Phantom Limb Pain; Peripheral Vascular Diseases
Keywords: transcutaneous electrical nerve stimulation
MeSH Terms: conditions — Phantom Limb; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TENS INTERVENTION (Active Comparator): In the immediately postoperative of limb amputation, TENS will be use in this patients during 24 hours. The intensity of the impulse will be determined in a test carried out 3 days before surgery. The other parameters will be continuous, biphasic, compensated and symmetric impulse, frequency of 80 Hz, time impulse between 250 and 290 microseconds, modulation time 5´´
  Interventions: Device: TENS INTERVENTION
- TENS NO INTERVENTION (Placebo Comparator): In the immediately postoperative of limb amputation, TENS will be use in this patients during 24 hours, but in this case TENS just will be on. No intensity impulse should be programmed.

INTERVENTIONS:
Device: TENS INTERVENTION — 24 hours of TENS treatment in the immediately postoperative of limb amputation
  Arms: TENS INTERVENTION

SUMMARY:
A growing body of literature indicates that up to 80% of amputees may have phantom limb pain (PLP). The first cause for limb loss is vascular disease. Usually, amputees who suffer from PLP are suboptimal treated. Therefore, many amputees are disabled by their chronic pain. The etiology and pathophysiology of PLP are poorly understood. Some studies suggest a somatosensory cortex reorganization. Transcutaneous Electrical Nerve Stimulation (TENS) is a analgesic technique. TENS apply a low voltage electrical current through the skin using surface electrodes in order to stimulate afferent nerve fibbers. Because of the lack of evidence to support any treatment for PLP, interest has turned to preventing it instead.

The aim of this study is to assess if the early use of TENS in the immediately postoperative of major limb amputation due to peripheral vascular disease, should decrease the PLP incidence. TENS should interfere in the mechanism of PLP production to level of the pain fibers conduction.

DETAILED DESCRIPTION:
Introduction:

Postamputation pain is highly prevalent after vascular limb amputation. The physiopathological basis should be divided in supraspinal, spinal and peripheral mechanisms. Supraspinal mechanism involve somatosensory cortical reorganization; spinal reorganization in the dorsal horn, occurs after deafferentation from peripheral nerve injury and peripherical nerve injury begins with the nerve section in surgery. All this factors seems to end into a somatosensory cortex reorganization. In this sense, it seems that our ability to prevent PLP depend on the capability to modulate the plasticity of the Central Nervous System (CNS).

Transcutaneous electrical nerve stimulation it´s a safe, easy and inexpensive analgesic technique acting on the conduction pathways of pain. An adequated program is mandatory: balanced symmetrical biphasic pulse, pulse length greater than 250microsg, modulated high frequency and electrodes placed over the dermatomes corresponding to lumbar-sacral spine; will be used in the intervention patients

Hypothesis:

In patients with TENS use during the immediately postoperative of major limb amputation due to peripheral vascular disease, phantom limb pain will appear with less frequency than in control patients.

Study population:

Patients undergoing major limb amputation for peripheral vascular disease.

Study design:

A randomized, prospective, blinded (patient, physician, statistician),clinical trial placebo versus intervention group study has been design.

In the intervention arm, TENS should be applied during the 24 hours immediately after limb amputation. The placebo arm, also will carry TENS but without an active program.

All patients should receive the standard analgesic treatment for limb amputation during their hospitalization time.

Evaluation and objectives:

Before surgery all patients made two test for pain evaluation: The Analogical Visual Scale and the DN4 questionnaire for neuropathic pain.

At 3 days, 1 month and 3 months after surgery, all patients will be evaluated about their pain using the recommended test for neuropathic pain:The Analogical Visual Scale and the DN4 (neuropathic pain 4) questionnaire for neuropathic pain . Also, at month 1 and 3th, two more test should be done in order to evaluate quality of life: The SF-12 (short form-12) health survey questionnaire about health and the Medical Outcomes Study (MOS) for sleep test.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years of both genders
* Critical limb ischemia (arteriopathic or diabetic aetiology)
* "MINI MENTAL TEST" (minimum 24 points)

Exclusion Criteria:

* Pace marker
* Don´t speak Spanish
* Not agreement with the study
* Dermatological lesion affecting the electrode place

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-11 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
PREOPERATIVE PAIN EVALUATION | 3 days before intervention
  Analogical Visual Scale: the patient indicate its pain level in the scale witch has an interval between 0-10 DN4 Test ( for neurophatic pain). This is the recommended test of the Spanish association on Anesthesiology for determinate neurophatic pain.
PREOPERATIVE NEUROPAThIC PAIN EVALUATION | 3 days before intervention
  DN4 Test ( for neuropathic pain). This is the recommended test of the Spanish association on Anesthesiology for determinate neuropathic pain. It consist in several questions to evaluate the clinical situation and some others about the physical situation.

SECONDARY OUTCOMES:
INMEDIATELY POSTOPERATIVE PAIN EVALUATION | 3 days after intervention
  Analogical Visual Scale: the patient indicate its pain level in the scale witch has an interval between 0-10
INMEDIATELY POSTOPERATIVE PAIN EVALUATION | 3 days after intervention
  DN4 Test ( for neuropathic pain). This is the recommended test of the Spanish association on Anesthesiology for determinate neuropathic pain. It consist in several questions to evaluate the clinical situation and some others about the physical situation.
1 MONTH POSTOPERATIVE PAIN EVALUATION | 1 MONTH
  Analogical Visual Scale: the patient indicate its pain level in the scale witch has an interval between 0-10
1 MONTH POSTOPERATIVE PAIN EVALUATION | 1 MONTH
  DN4 Test ( for neuropathic pain). This is the recommended test of the Spanish association on Anesthesiology for determinate neuropathic pain. It consist in several questions to evaluate the clinical situation and some others about the physical situation.
1 MONTH POSTOPERATIVE HEALTH EVALUATION | 1 MONTH
  Test SF-12 about health situation. This is the recommended test of the Spanish Pain society for subjective evaluation of health situations. It consist in 12 questions about its own perceptions, employment status, daily activities, frame of mind
1 MONTH POSTOPERATIVE SLEEP EVALUATION | 1 MONTH
  Test MOS (Sleep Scale from the Medical Outcomes Study) Some questions for sleep evaluation
3 MONTH POSTOPERATIVE PAIN EVALUATION | 3 MONTH
  Analogical Visual Scale: the patient indicate its pain level in the scale witch has an interval between 0-10
3 MONTH POSTOPERATIVE PAIN EVALUATION | 3 MONTH
  DN4 Test ( for neuropathic pain). This is the recommended test of the Spanish association on Anesthesiology for determinate neuropathic pain. It consist in several questions to evaluate the clinical situation and some others about the physical situation.
3 MONTH POSTOPERATIVE HEALTH EVALUATION | 3 MONTH
  Test SF-12 about health situation. This is the recommended test of the Spanish Pain society for subjective evaluation of health situations. It consist in 12 questions about its own perceptions, employment status, daily activities, frame of mind
3 MONTH POSTOPERATIVE SLEEP EVALUATION | 3 MONTH
  Test MOS (Sleep Scale from the Medical Outcomes Study) Some questions for sleep evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Bodega, Mrs, Principal Investigator — Hospital General Universitario de Castellon. Avenida Benicassim sn 12004. Castellon. Spain
Locations (1):
- hospital General Universitario de Castellon, Castellon, Castellon de La Plana, Spain